CLINICAL TRIAL: NCT01654289
Title: Meditation or Exercise for Preventing Acute Respiratory Infection (MEPARI-2)
Brief Title: University of Wisconsin Meditation & Exercise Cold Study
Acronym: MEPARI-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-0207; R01AT006970 (NIH)
Record Dates: First submitted 2012-07-19; First posted 2012-07-31 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Acute Respiratory Infection
Keywords: respiratory tract infections; common cold; exercise; influenza; meditation
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold; Motor Activity; Influenza, Human | interventions — Mindfulness; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mindfulness Meditation (Experimental): Training will consist of a standardized 8-week Mindfulness Based Stress Reduction (MBSR) program, including 2½ hour weekly sessions and approximately 45 minutes per day at-home daily practice.
  Interventions: Other: Mindfulness Meditation
- Exercise (Experimental): The exercise intervention structure is consistent with many standardized exercise programs. The exercise program will match the meditation program in duration (8 weeks), attention (weekly 2½ hour group sessions), and intensity (daily 45 minute at-home practice).
  Interventions: Other: Exercise
- Wait-list control (No Intervention): Apart from not attending any of the specific meditation or exercise training sessions, those in the control group will be treated in essentially the same manner as "experimental" participants.

INTERVENTIONS:
Other: Mindfulness Meditation — Training will consist of a standardized 8-week Mindfulness Based Stress Reduction (MBSR) program, including 2½ hour weekly sessions and regular at-home daily practice. Didactic sessions center on awareness of physical, emotional, cognitive, and interpersonal responses to stress. A half day meditation "retreat" on a weekend day at the end of week 6 will allow participants to practice their skills.
  Other Names: MBSR
  Arms: Mindfulness Meditation
Other: Exercise — Exercise training will primarily focus on walking or jogging, activities that are convenient, easy to teach and do not require special equipment. Individualized programs will be developed for those who have access to specific equipment, are unable to do walking/jogging, or prefer different types of exercise. Each weekly exercise session will include 1½ hours of didactic and 1 hour of group exercise. A half day exercise retreat designed to match the meditation retreat will occur the weekend of week 6. The retreat will include didactics, group discussion and activities, and individualized exercise practice.
  Other Names: physical activity
  Arms: Exercise

SUMMARY:
The primary goal of this project is to determine whether behavioral training in mindfulness meditation or moderate intensity sustained exercise will lead to reductions in acute respiratory infection (ARI) illness, such as common cold and influenza like illness. Specifically, this project aims to:

1. Determine whether an 8-week training program in mindfulness meditation, as compared to the control group, will lead to significant reductions in incidence, duration, and severity of ARI illness.
2. Determine whether an 8-week training program in moderate intensity sustained exercise, as compared to the control group, will lead to reductions in incidence, duration, and severity of ARI illness.
3. Assess whether any observed reductions in ARI illness are accompanied by fewer ARI-related health care visits and less time lost to productive work (reduced absenteeism).
4. Compare the potential benefits of mindfulness meditation to those from moderate intensity sustained exercise.
5. Discern potential mediating factors and causal pathways that might help explain how these interventions lead to improved ARI illness-related outcomes.

The investigators' preliminary findings suggest substantial benefit of these interventions in terms of reduced incidence, duration and severity of ARI illness, with corresponding reductions in days of work lost to illness. If the proposed research confirms these findings, there will be major implications for public and private health-related policy and practice, as well as for scientific knowledge regarding health maintenance and disease prevention.

DETAILED DESCRIPTION:
Acute respiratory infection (ARI), including common cold and influenza, is a leading cause of morbidity and mortality, and has a major economic impact. Both mental and physical health are linked to ARI burden. For example, people who report more negative emotion and higher stress are more likely to get ARI. Exercise affects the immune system, improves physical and mental health, and may protect against ARI illness. Mindfulness meditation reduces perceived stress, influences the immune system, and may protect against ARI. The investigators' own recent NCCAM-funded trial randomized 154 people to 3 groups: 1) meditation, 2) moderate intensity exercise, or 3) wait-list control. For the 149 people followed to study completion, there were 40 ARI episodes and 453 days of illness in the control group, 27 episodes and 257 days of ARI illness in the meditation group, and 26 episodes and 241 days of ARI illness in the exercise group. Corresponding reductions in ARI-related work days lost to ARI illness were observed. The proposed research will build upon these findings with refined methodology in a larger sample to: A) determine whether these findings are replicable, and B) investigate potential explanatory pathways.

This research will use state-of-the-art randomized controlled trial (RCT) methodology to assess potential effects of meditation or exercise on ARI outcomes. This will be a 5-year project, with 4 yearly cohorts of n=99 per cohort randomized into 3 groups of n=33 each. Assuming 9% loss to follow-up, the final sample size will be n=360 study participants, with n=120 in each comparison group. Participants will be randomized to 1 of 3 groups: 1) an 8-week training program in mindfulness meditation, 2) an attention, duration and location-matched program in progressive exercise, or 3) a non-interventional wait-list control group. Each cohort will be observed for 8 months comprising the annual cold and flu season. Enrollment, randomization and study interventions will begin in September of each year. Participants will be monitored by weekly self-report through May. Summers will be used for data cleaning, preliminary analyses, and for recruiting the next year's cohort.

The primary goal of this project is to determine whether behavioral training in mindfulness meditation or moderate intensity sustained exercise can lead to reductions in acute respiratory infection (ARI) illness, such as common cold and influenza like illness. The primary outcome will be severity-weighted total days of ARI illness (global severity), calculated as trapezoidal approximation to area under the time severity curve during ARI illness, with severity assessed once daily using self-reports on the validated Wisconsin Upper Respiratory Symptom Survey (WURSS-24).

Computer-assisted weekly monitoring will assure that ARI illness episodes are detected, and will serve to document secondary outcomes, including health care utilization and work or school absenteeism. Visits to health care facilities and time lost from work and school will be documented, then classified as ARI-related (or not) by personnel blinded to allocation. Questionnaire measures assessing perceived stress, self-efficacy, sleep quality, depression, and general mental and physical health will also be analyzed as secondary outcomes. Degree of stress reduction, mindfulness, positive and negative emotion, social support, self-efficacy and sleep quality will be analyzed as potential mediators of effects of interventions on outcomes.

Laboratory assessed objective measures will primarily serve to corroborate self-reports of disease severity, but will also be analyzed as potential mediators of effects of behavioral interventions on ARI illness incidence, duration, and severity. As potential mediators, pro-inflammatory cytokines (CRP, IL-6, IL-8, IP-10) will be assessed as change from baseline to one month after the 8 week behavioral interventions finish. These will serve as indicators of a pro-inflammatory state. Repeating these assays 3 months later will assess whether pro-inflammatory changes from baseline will be sustained. Cytokines from samples taken during ARI illness will be assessed as corroborating biomarkers of disease severity. Identification of viral agents using multiplex PCR will also serve to corroborate ARI self-reports.

Self-report measures of perceived stress, positive and negative emotion, self-efficacy, social support, sleep quality, mindfulness, and general mental and physical health will be used to assess potential pathways through which interventions may exert influence on primary outcomes. Potential mediating effects of psychological and physical health domains will be assessed using appropriate mediation (process) analysis statistical models.

Primary efficacy analysis will contrast total days of illness and area-under-curve global severity in each intervention group with corresponding values in the control group. Unadjusted contrasts will be done by t-test, using variable transformation if skewness requires. Adjusted analyses will be based on zero-inflated regression models taking into account the episodic and variable nature of ARI illness. Zero-inflated regression models incorporate a logistic sub-model to account for people without ARI illness, and a linear sub-model to account for the variability in continuous measures of severity and duration. These will employ conservative estimates with standard error inflated using Huber/White maximum likelihood estimation. Co-variates to be controlled for in this model will include: age, sex, body mass index, smoking status, comorbidity, highest level of education achieved, neuroticism, conscientiousness, general physical health and general mental health. The null hypotheses of "no effect on primary outcome" will be rejected in favor of alternative hypothesis of "some effect" if p-values are ≤0.025. Confidence intervals will be constructed for all outcome variables, allowing estimation of effect size. Zero-inflated regression models for primary efficacy analyses will be done using M-Plus version 6.1or similar software.

Influence of interventions on secondary outcomes will be assessed using ANOVA-based multivariate regression models using SAS software. Adjustment for multiple comparisons will be incorporated, and interpretation will be cautious. In general, the investigators' will want to see relationships with p<0.01 in order to justify tentative null hypothesis rejection. Pre-planned secondary efficacy analyses will include effects of interventions on: 1) absenteeism, 2) health care utilization, 3) general physical health (SF-12), 4) general mental health (SF-12); 5) perceived stress (PSS-10), 6) self-efficacy (MSES, ESE), 7) sleep quality (PSQI), 8) body weight (BMI), 9) blood pressure and 10) pro-inflammatory cytokines. One-sided testing will be based on the underlying hypotheses that the behavioral trainings lead to improved physical and mental health, sleep quality and self-efficacy, and to reductions in absenteeism, health care utilization, stress, body weight, blood pressure and proinflammatory cytokines.

Apart from flu shots, hand-washing, smoke avoidance, and maintenance of general health, there are no known safe and effective prevention strategies for acute viral respiratory infection. Interventions to be tested are low risk, and more likely to confer benefit than harm. Influenza vaccination (flu shots) will be provided free of charge to all participants, and could be considered a benefit. Participants will not be required to forego any proven or accepted preventions or treatments, and in fact will be encouraged to seek appropriate medical attention for any condition, including respiratory infection, and to continue their regular health care practices. Antibiotics, anti-influenza antivirals, and other ARI treatments will not be disallowed, but instead will be tracked as secondary outcomes. In general, participants will be asked to continue the study interventions they are assigned, and to forego the study interventions they are not assigned. However, they will be informed that they remain free to make their own health care, behavioral and life style decisions. In particular, exercise will not be discouraged for participants in the meditation or wait-list control group, as exercise is known to confer some health benefit. However, the investigators' will ask participants in the exercise and control group to refrain from starting a meditation program, and that all participants refrain from starting any purportedly immune-modifying supplements (eg, echinacea, ginseng, zinc, elderberry, etc.), unless advised to do so by their physicians. If any participants do choose to actively begin an intervention they were not assigned (i.e. a person randomized to exercise chooses to take the mindfulness meditation course instead), the investigators' will ask them to continue in the study, and will use that "cross-over" information in secondary analyses using the principles outlined in Section 4.3 of the protocol.

This proposed study was submitted to and approved by the Human Subjects Committee of the Health Sciences Institutional Review Board of the University of Wisconsin - Madison (UW HS-IRB), and will be in compliance with HIPAA and all other federally mandated human subjects regulations. All members of the research team will complete the protection of human subjects' tutorial required by the UW HS-IRB's Human Subjects Committee prior to the study's initiation. All named UW Co-Investigators, Consultants, and current Project Personnel have in fact already completed this tutorial. All study personnel, including research assistants, will be trained in confidentiality, informed consent procedures, and other aspects of human subject protection.

A Data and Safety Monitoring Committee (DSMC) will oversee human subjects recruitment and monitoring, and will function independently of the principal investigator and co-investigators. The investigators' expect that this committee will function similarly to that established for the first MEPARI trial, and will choose to meet once or twice yearly to monitor recruitment and retention, and to provide oversight and guidance in relation to safety, bioethics, and other human subjects concerns that may arise.

Acute infection from influenza and other respiratory viruses leads to much human suffering and loss of economic productivity. The investigators' own evidence suggests that training in either meditation or exercise may lead to substantial reductions in ARI disease burden and work absenteeism. In addition to testing whether the investigators' findings are replicable in a larger sample with refined methodology, this proposed comparative effectiveness translational research will investigate mechanisms of action and provide initial estimates of cost-effectiveness. If positive findings are confirmed, this line of research could have direct and immediate impact on public and private health-related policies and clinical practice, as well as on scientific understanding of respiratory infection.

A copy of the full protocol (including references) is available upon request.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-69 years at study entry.
* Must answer "Yes" to either "Have you had at least 2 colds in the last 12 months?" and/or "On average do you get at least 1 cold per year?"
* Prospective participants must meet the American Heart Association guidelines for suitability for an exercise program. Prospective participants will be advised (but not required) to seek their physicians' advice before enrollment.
* Self-reported ability and willingness to follow through with either exercise or meditation training, or neither, according to randomized allocation, and to participate in blood draws, nasal wash, self-report questionnaires, and weekly monitoring for 9 months.
* A score of 14 or lower on the PHQ-9 depression screen, self-reported both at entrance to run-in trial and again just prior to enrollment in the main study.
* Fluency and literacy in English language sufficient for understanding the study protocol and completing questionnaires.
* Successful completion of tasks during run-in period, including 2 in-person appointments, 1 phone contact, 1 set of homework questionnaires, and baseline nasal wash and blood draw.

Exclusion Criteria:

* Current or recent use of meditative practice, or previous meditation training. Assessed by answering "Yes" to any of the following questions: Do you meditate on a regular basis? In the last year, have you meditated at least weekly for 2 or more months in a row? Have you ever been trained in meditation? Have you ever been involved in a mindfulness class or mindfulness practice?
* Potential participants must not engage in moderate exercise more than twice per week or vigorous exercise more than once per week, as assessed by the following questions adapted from the Behavioral Risk Factor Surveillance System (BRFSS) classification system: On average, how many times per week do you engage in moderate recreational activities such as walking, tennis doubles, ballroom dancing, weight training, or similar activities that last at least 20 minutes per occasion? A) Less than 1 time per week; B) 1 time per week; C) 2 times per week; D) 3 times per week; E) >4 times per week. How many times per week do you engage in vigorous sport and recreational activities such as jogging, swimming, cycling, singles tennis, aerobic dance or other similar activities lasting at least 20 minutes per occasion? A) Less than 1 time per week; B) 1 time per week; C) 2 times per week; D) 3 or more times per week.
* Women who are pregnant at screening or plan to become pregnant during the course of the study (determined by self-report) will be excluded. Women who become pregnant any time during the course of the trial will not be dropped and will continue to be followed throughout the duration of the study.
* Physical, medical or mental condition(s) precluding adherence to study protocol. Conditions include: malignant disease (prospective participants' physicians to advise and Dr. Barrett, and/or designee Dr. Rakel or Dr. Muller, to make final decision); and function-impairing psychopathology (prospective participants' psychiatrist or psychologist to advise). Questionable cases will be reviewed by the study physicians.
* True contraindication for influenza vaccine (flu shots) or refusal to accept influenza vaccine. Subjects will be asked to verify they have a) no known egg allergy, b) no prior reaction to influenza vaccine, and c) never been told they have Guillain-Barre Syndrome.
* Current use or forecasted need for immunoactive drugs (eg. steroids, immunosuppressants, chemotherapy); nonsteroidal antiinflammatories will be allowed.
* Immune deficiency or auto-immune disease (eg. HIV/AIDS, lupus, rheumatoid arthritis, multiple sclerosis, inflammatory bowel disease). Questionable cases will be reviewed by study physicians.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2012-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barrett, MD PhD, Principal Investigator — University of Wisconsin Department of Family Medicine
Locations (1):
- University of Wisconsin Department of Family Medicine, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Meyer JD, Torres ER, Grabow ML, Zgierska AE, Teng HY, Coe CL, Barrett BP. Benefits of 8-wk Mindfulness-based Stress Reduction or Aerobic Training on Seasonal Declines in Physical Activity. Med Sci Sports Exerc. 2018 Sep;50(9):1850-1858. doi: 10.1249/MSS.0000000000001636. PMID 30113538
- [Derived] Barrett B, Hayney MS, Muller D, Rakel D, Brown R, Zgierska AE, Barlow S, Hayer S, Barnet JH, Torres ER, Coe CL. Meditation or exercise for preventing acute respiratory infection (MEPARI-2): A randomized controlled trial. PLoS One. 2018 Jun 22;13(6):e0197778. doi: 10.1371/journal.pone.0197778. eCollection 2018. PMID 29933369
- [Derived] Goldstein E, Topitzes J, Brown RL, Barrett B. Mediational pathways of meditation and exercise on mental health and perceived stress: A randomized controlled trial. J Health Psychol. 2020 Oct;25(12):1816-1830. doi: 10.1177/1359105318772608. Epub 2018 May 7. PMID 29733230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from the greater Madison WI (USA) community between July 2012 and September 2016.
Pre-assignment Details: Prospective subjects were met in person for informed consent and enrollment in a 2-week run-in trial. Run-in tasks included baseline questionnaires, at least one phone contact, self-report questionnaires at home, and a follow-up in-person appointment. Successful completion of run-in activities allowed participants to enroll in main study.
Period: Overall Study
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Started | 138 | 137 | 138
Completed | 111 | 109 | 133
Not Completed | 27 | 28 | 5
Not completed — Withdrawal by Subject | 10 | 8 | 5
Not completed — Withdrew from intervention only | 17 | 20 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control | Total
Number analyzed (Participants) | 138 | 137 | 138 | 413
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.4) | 49.2 (11.2) | 50.7 (12.1) | 49.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 107 | 101 | 313
  Male | 33 | 30 | 37 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 5 | 8 | 24
  Not Hispanic or Latino | 127 | 132 | 130 | 389
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 8 | 3 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 14 | 6 | 25
  White | 121 | 105 | 123 | 349
  More than one race | 7 | 10 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 138 | 137 | 138 | 413

OUTCOME MEASURES:

1. Primary Outcome: Severity-weighted Total Days of ARI Illness
Description: The primary outcome will be severity-weighted total cumulative days of ARI illness (global severity), calculated as trapezoidal approximation to area under the time severity curve during ARI illness, with severity assessed once daily using self-reports on the validated Wisconsin Upper Respiratory Symptom Survey (WURSS-24). Incidence (number of ARI episodes in each group) and duration (total number of days of ARI illness) are components of the primary outcome, and will be analyzed separately.
Time Frame: 8 months
Measure: Number; unit: severity*days
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
severity*days | 1045 | 1010 | 1210

2. Secondary Outcome: Absenteeism
Description: Employment, including type of work, hours per week worked, and compensation, assessed as hourly wage, will be assessed at enrollment. Each week throughout the study participants will complete questions to assess number of hours of work missed. Study personnel blinded to allocation group status will assess and classify reasons for missed work as either ARI-related or not ARI-related. Presented as a total cumulative number of days missed of work due to an ARI-related event.
Time Frame: 8 months
Measure: Number; unit: Total # of ARI-related Missed Work days
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
Total # of ARI-related Missed Work days | 73 | 81 | 105

3. Secondary Outcome: Health Care Utilization
Description: Cumulative total number of health care visits, ARI-related health care visits, and ARI-related prescriptions, including antibiotics and anti-influenza anti-virals will be documented. Each weekly communication will include the question, "Have you seen a doctor or visited a clinic, hospital or urgent care center?" Persons answering "Yes" will be asked the reason for the visit. Those answers will then be classified by blinded study personnel as either "Related," or "Unrelated" to ARI illness, including upper respiratory infection, influenza, pharyngitis, acute sinusitis, bronchitis, and pneumonia.
Time Frame: 8 months
Measure: Number; unit: Total # ARI-related Medical visits
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
Total # ARI-related Medical visits | 22 | 21 | 24

4. Secondary Outcome: SF-12
Description: Also known as the Medical Outcomes Study Short Form, this 12-item questionnaire is commonly used to measure overall health, including physical (SF12-P) and mental health (SF12-M) subscales. It has been extensively assessed for reliability, responsiveness and criterion validity. In this study, it will be used to assess potential changes in general physical and mental health due to interventions, and as a covariate to control for baseline between-person differences in multivariate efficacy analyses. Physical and Mental Health Composite Scores are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline and 8 months (exit from study)
Population: Obtained participant data reported.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
score on a scale
  SF12-P Baseline | 51.2 [35.6 to 67.1] | 51.4 [34.9 to 67.8] | 51.4 [35.1 to 67.6]
  SF-12-P Exit: number analyzed (Participants) | 129 | 129 | 129
  SF-12-P Exit | 50.5 [31.4 to 71.7] | 51.9 [32.2 to 70.9] | 51.5 [33.9 to 69.2]
  SF12-M Baseline | 48.0 [28.0 to 67.1] | 47.9 [27.1 to 68.0] | 47.6 [28.2 to 66.9]
  SF-12-M Exit: number analyzed (Participants) | 128 | 129 | 132
  SF-12-M Exit | 49.7 [25.2 to 66.5] | 47.8 [26.2 to 65.6] | 45.9 [25.1 to 66.6]

5. Secondary Outcome: Perceived Stress Scale (PSS-10)
Description: The PSS-10 has been validated in multiple studies. PSS scores predict rates of viral infection among volunteers inoculated with rhinovirus, and correlate with physiologic and self-report indicators of ARI illness, including nasal IL-6 level. Because stress reduction is one of the hypothesized mechanisms of action, this study population will include working-age participants, who are presumed to be more stressed. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
Time Frame: Baseline and 8 months (exit from study)
Population: Obtained participant data reported.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
score on a scale
  PSS-10 Baseline | 13.1 [-0.3 to 25.0] | 13.3 [-0.5 to 25.3] | 12.4 [0.8 to 24.0]
  PSS-10 Exit: number analyzed (Participants) | 128 | 129 | 133
  PSS-10 Exit | 11.6 [0.8 to 26] | 13.3 [-0.5 to 27.4] | 13.4 [0.6 to 26.2]

6. Secondary Outcome: Mindfulness-based Self Efficacy Scale (MSES)
Description: The MSES is one of the more recent questionnaires, developed by Cayoun and Freestun to assess effects of MBSR training on perceived self-efficacy. The MSES assesses 7 domains related to mindfulness self-efficacy, including behavior, cognition, interoception, affect, interpersonal, avoidance and mindfulness. The MSES will provide a nice counterpart to the ESES to help distinguish effects of interventions on ARI outcomes. The lower the score, the lower self-efficacy is in using mindfulness skills.
  The current lack of psychometric data for the MSES renders the following ranges very tentative. They are currently only a rough clinical guide and scores must be interpreted with caution.
  0-34 Poor sense of self-efficacy 35-69 Weak sense of self-efficacy 70-104 Moderate sense of self-efficacy 105-140 Good sense of self-efficacy
Time Frame: 8 months (exit from study)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
score on a scale | 97.6 (15.7) | 97.3 (14.7) | 96.8 (14.6)

7. Secondary Outcome: Exercise Self-Efficacy Scale (ESES)
Description: Self-efficacy has been defined as "the belief in one's capabilities to organize and execute the courses of action required to manage prospective situations." The ESES scale was developed based on work by Bandura and colleagues,and has been validated by Shin, Kroll,and Everett. For this study, the ESES will be used to verify results of the exercise intervention, and to help explain potential mediational effects of exercise. The total score is derived by summing the scores for the individual items; possible scores range from 0 to 180. Total score (out of 180) is sum of item scores. Higher score represents greater perceived self efficacy.
Time Frame: Baseline and 8 months (exit from study)
Population: Obtained participant data reported.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
score on a scale
  ESES - Baseline: number analyzed (Participants) | 138 | 136 | 137
  ESES - Baseline | 112.5 [41.0 to 191.0] | 112.4 [40.3 to 191.6] | 116.0 [39.9 to 192.1]
  ESES - Exit: number analyzed (Participants) | 128 | 129 | 138
  ESES - Exit | 94.3 [8.9 to 160.2] | 104.4 [13.4 to 155.8] | 84.6 [13.3 to 155.9]

8. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Sleep quality has been linked to several important quality of life and health outcomes. The PSQI is widely used and has been assessed for reliability and validity.In this study, improved sleep is a potential mediator of intervention effects, and a potentially important outcome on its own. The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Time Frame: Baseline and 8 months (exit from study)
Population: Obtained participant data reported.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
score on a scale
  PSQI - BASELINE: number analyzed (Participants) | 136 | 133 | 136
  PSQI - BASELINE | 5.8 [-0.7 to 12.0] | 6.2 [-1.4 to 12.7] | 5.7 [-0.8 to 12.1]
  PSQI - EXIT: number analyzed (Participants) | 128 | 127 | 132
  PSQI - EXIT | 5.1 [-0.1 to 11.8] | 5.3 [-0.4 to 12.0] | 5.8 [-1.3 to 13.0]

9. Secondary Outcome: Body Mass Index (BMI)
Description: Body habitus is associated with many disease processes, and may be related to immune function and susceptibility to respiratory infection. Height will be assessed at baseline only. Weight will be measured at baseline, 1 and 4 months post-intervention, and at exit. Baseline BMI will be calculated and used as a covariate in statistical models. BMI will also be considered a secondary outcome of potential importance.
Time Frame: Baseline and 8 months (exit from study)
Population: Obtained participant data reported.
Measure: Mean (Full Range); unit: kg/m2
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
kg/m2
  BMI - BASELINE | 29.8 [13.7 to 44.4] | 29.3 [15.4 to 42.7] | 29.0 [16.0 to 42.0]
  BMI - EXIT: number analyzed (Participants) | 128 | 128 | 132
  BMI - EXIT | 28.2 [24.2 to 33.4] | 27.4 [24.3 to 32.0] | 27.9 [24.1 to 33.0]

10. Secondary Outcome: Blood Pressure
Description: Standard brachial blood pressure will be assessed by trained nurses using calibrated sphygmomanometers.
Time Frame: Baseline and 8 months (exit from study)
Population: Obtained participant data reported.
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
mm Hg
  Systolic - Baseline | 120.4 [92.0 to 156.4] | 121.8 [94.2 to 154.2] | 124.2 [91.6 to 156.8]
  Diastolic-Baseline | 74.3 [59.4 to 92.3] | 75.0 [58.3 to 93.4] | 75.8 [57.7 to 94.0]
  Systolic - Exit: number analyzed (Participants) | 127 | 127 | 131
  Systolic - Exit | 121.0 [109.0 to 133.0] | 122.0 [108.0 to 130.0] | 124.0 [113.0 to 132.0]
  Diastolic - Exit: number analyzed (Participants) | 127 | 127 | 131
  Diastolic - Exit | 77.0 [69.0 to 82.0] | 76.0 [69.0 to 82.0] | 78.0 [71.0 to 83.0]

11. Secondary Outcome: Pro-Inflammatory Cytokines
Description: Laboratory-assessed objective measures will primarily serve to corroborate self-reports of disease severity. High sensitivity C-reactive protein (HS-CRP) is a well-established indicator of disease severity during respiratory infection, and can be measured in serum and in nasal wash.Concentrations of interleukin-6 (IL-6)and interleukin-8 (IL-8)in nasal wash have been shown to correlate with illness severity. More recently, interferon-gamma-induced protein 10 (IP-10) has been shown to be measurably increased in both serum and nasal wash during times of acute viral ARI. Biomarker levels were measured at the two standardized follow-up visits in December and March when participants were not ill.
Time Frame: Baseline, 4 months post-intervention (December) and 8 months post-intervention (March).
Population: Obtained participant data reported.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
Number analyzed (Participants) | 138 | 137 | 138
pg/mL
  hsCRP - Baseline | 1.6 [0.7 to 4.5] | 1.4 [0.6 to 3.9] | 1.5 [0.7 to 4.8]
  hsCRP - December: number analyzed (Participants) | 132 | 127 | 134
  hsCRP - December | 1.7 [0.8 to 4.8] | 1.7 [0.7 to 3.3] | 1.6 [0.7 to 4.4]
  hsCRP - March: number analyzed (Participants) | 127 | 126 | 131
  hsCRP - March | 1.3 [0.7 to 3.3] | 1.3 [0.6 to 3.2] | 1.4 [0.6 to 3.9]
  IL-6 nasal - Baseline: number analyzed (Participants) | 133 | 129 | 132
  IL-6 nasal - Baseline | 1.3 [0.8 to 2.2] | 1.0 [0.6 to 2.1] | 1.1 [0.5 to 2.3]
  IL-6 nasal - December | 1.7 [0.8 to 3.9] | 1.8 [0.8 to 2.9] | 1.3 [0.6 to 2.8]
  IL-6 nasal - March: number analyzed (Participants) | 128 | 129 | 130
  IL-6 nasal - March | 1.6 [0.9 to 2.6] | 1.6 [0.8 to 2.8] | 1.6 [0.8 to 3.6]
  IL-6 serum - Baseline | 1.6 [1.0 to 2.8] | 1.8 [1.1 to 2.9] | 1.7 [1.0 to 2.9]
  IL-6 serum - December: number analyzed (Participants) | 132 | 128 | 134
  IL-6 serum - December | 1.6 [0.9 to 3.2] | 1.7 [1.0 to 3.0] | 1.5 [1.0 to 2.6]
  IL-6 serum - March: number analyzed (Participants) | 127 | 127 | 132
  IL-6 serum - March | 1.7 [0.9 to 2.6] | 1.6 [0.9 to 2.5] | 1.8 [1.1 to 3.0]
  IP-10 - Baseline | 141 [117 to 183] | 156 [126 to 198] | 152 [127 to 198]
  IP-10 - December: number analyzed (Participants) | 132 | 128 | 134
  IP-10 - December | 140 [116 to 183] | 139 [116 to 172] | 148 [121 to 205]
  IP-10 - March: number analyzed (Participants) | 127 | 126 | 132
  IP-10 - March | 149 [114 to 192] | 145 [111 to 190] | 147 [123 to 192]
  IL-8 - Baseline | 167 [86 to 313] | 157 [79 to 271] | 194 [87 to 352]
  IL-8 - December: number analyzed (Participants) | 133 | 129 | 132
  IL-8 - December | 238 [144 to 356] | 214 [127 to 354] | 255 [140 to 446]
  IL-8 - March: number analyzed (Participants) | 128 | 129 | 130
  IL-8 - March | 258 [157 to 424] | 227 [158 to 414] | 248 [155 to 390]

ADVERSE EVENTS:
Time Frame: Each cohort was followed for no more than 10 months (August through June).
Arm/Group | Mindfulness Meditation | Exercise | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/137 | 0/138
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/137 | 0/138
Other Adverse Events (participants affected / at risk) | 10/138 | 20/137 | 16/138
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Meditation (N=138) | Exercise (N=137) | Wait-list Control (N=138)
Cardiac Disorders (Cardiac disorders) | 1 (1) | 8 (8) | 1 (1)
General (General disorders) | 5 (5) | 7 (7) | 8 (8)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 10 (10) | 13 (13) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT01654289/Prot_SAP_000.pdf